CLINICAL TRIAL: NCT00227357
Title: SPNS - An Evaluation of Innovative Methods for Integrating Buprenorphine Opioid Abuse Treatment in HIV Primary Care
Brief Title: The CORE Buprenorphine Project - An HIV Primary Care Program Demonstration
Acronym: BUP
Status: Completed | Type: Observational
Sponsor: Ruth M. Rothstein CORE Center (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); The New York Academy of Medicine (Other)
Responsible Party: Jeffrey D. Watts, M.D., The Ruth M. Rothstein CORE Center
Other Study IDs: 1-H97HA03796-01-00
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections; AIDS; Opiate Dependence; Post-Traumatic Stress Disorders
Keywords: HIV; AIDS; Buprenorphine; Methadone; Primary care; dual diagnosis; ptsd
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Opioid-Related Disorders; Stress Disorders, Post-Traumatic | interventions — Naloxone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Buprenorphine: Study patients receiving buprenorphine treatment
  Interventions: Drug: On-site - buprenorphine/naloxone (Suboxone)
- Comparison: Study patients receiving methadone or no agonist treatment
  Interventions: Drug: Off-site - methadone or no agonist

INTERVENTIONS:
Drug: On-site - buprenorphine/naloxone (Suboxone) — Tablet, sub-lingual, 8/2 mg, 1-3 daily
  Groups: Buprenorphine
Drug: Off-site - methadone or no agonist
  Groups: Comparison

SUMMARY:
The goal of this study is to develop and evaluate an innovative model of care to better serve patients who are both HIV-infected and opioid-dependent.

DETAILED DESCRIPTION:
Hypothesis: HIV, opioid dependent patients provided agonist therapy at the site of their primary care will have better retention, utilization of services, health, social and quality of care measures and psychiatric treatment outcomes.

The Buprenorphine Project is an examination of two methods of service delivery. The purpose of this study is to assess the feasibility, cost and effectiveness of an intervention designed to integrate buprenorphine treatment for opioid dependence into HIV primary care at the CORE Center. For this project we will provide buprenorphine to 60 opioid dependent patients at any one time and will compare this on-site treatment group to 60 opioid dependent HIV+ patients who select off-site methadone or no agonist treatment at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patient of the CORE Center
* HIV-infected (confirmed by HIV assay results)
* Opioid-dependent (by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision [DSM-IV-TR] criteria)
* Fluent in English or Spanish
* Planning to stay in Chicago area for the next 12 months

Exclusion Criteria:

* Liver function tests (LFTs) (transaminase only) at 5 times or higher than normal
* DSM-IV-TR criteria for benzodiazepine abuse or dependence within the past 6 months
* DSM-IV-TR criteria for alcohol dependence within the past 6 months or actively suicidal
* Psychiatric impairment that impedes ability to consent
* Methadone dose exceeds level allowing for safe transition to buprenorphine
* Pregnant women or women actively trying to become pregnant
* Clinical judgement that patient is inappropriate for medical or psychiatric reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving buprenorphine treatment Patients not receiving buprenorphine treatment (methadone or none)
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D. Watts, M.D., Principal Investigator — The CORE Center and John H. Stroger, Jr. Hospital of Cook County, Affiliates of the Cook County Bureau of Health Services
Locations (1):
- The CORE Center, Chicago, Illinois, United States

REFERENCES:
- See also: Click here for more information about The CORE Center. — http://www.corecenter.org
- See also: Evaluation and Support Center for the Mult-site Buprenorphine Study — http://www.bhives.org